CLINICAL TRIAL: NCT02016755
Title: A Phase IIB Pilot Study to Confirm the Feasibility and Tolerability of a Modified Dosage Regimen of AMG0001 in Subjects With Critical Limb Ischemia
Brief Title: A Phase IIB Pilot Study of a Modified Dosage Regimen of AMG0001 in Subjects With Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG-CLI-0209
Record Dates: First submitted 2013-11-26; First posted 2013-12-20 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Critical Limb Ischemia; Vascular Diseases; Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Vascular Disease; CLI; Critical Limb Ischemia; PAD; AnGes; HGF Plasmid; HGF; Hepatocyte Growth Factor Plasmid; gene therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG0001 (Experimental): Hepatocyte Growth Factor (HGF) Plasmid
  Interventions: Biological: HGF Plasmid

INTERVENTIONS:
Biological: HGF Plasmid — Intramuscular injection in the affected limb.
  Other Names: AMG0001

SUMMARY:
The purpose of the study is to confirm the feasibility of study procedures and the tolerability of a new dose regimen of AMG0001 in subjects with Critical Limb Ischemia (CLI)

DETAILED DESCRIPTION:
The primary objectives of the study are:

1. To confirm the feasibility of study-related activities and the tolerability of a modified dosage regimen of AMG0001 in CLI
2. To evaluate safety of AMG0001

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stable CLI (Severe Rutherford 4 and Rutherford 5) who have no option for revascularization by endovascular intervention or surgical bypass or a poor option (high risk) for revascularization by surgery and no option for an endovascular intervention
* Subjects 40-90 years of either gender who have signed an informed consent
* Subjects currently are taking a statin and an anti-platelet agent
* If female, the subjects must not be of child bearing potential, e.g., post-menopausal or surgically sterile.
* If a male subject is of reproductive potential, he must agree to use an accepted and effective (barrier) form of birth control starting with the first dose of study product and continue for 12 weeks from the last dose of study product.
* Subjects with a previous medical history of myocardial infarction and/or stroke should have adequate management of risk factors to prevent secondary occurrence.
* Subjects should have the ability to understand the requirements of the protocol and agree to return for the required study visits and assessments

Exclusion Criteria:

* Subjects whose CLI status is unstable (spontaneous marked improvement or marked worsening during the screening period).
* Subjects who may require a major amputation (amputation at or above the ankle) within 4 weeks of Day 0 (± 4 weeks of Day 0).
* Subjects with ulcers with exposure of tendons, osteomyelitis or uncontrolled infection or with the largest ulcer that is greater than 20 cm2 in area (>10 cm2 area if on the heel).
* Subjects with purely neuropathic or venous ulcers.
* Subjects in Rutherford 6 class.
* Subjects who have had revascularization by surgery or angioplasty within 3 months, unless the procedure has failed based on the anatomy or the hemodynamic measurements.
* Subjects with a diagnosis of Buerger's disease (Thrombo-angiitis Obliterans).
* Subjects currently receiving immunosuppressive, chemo or radiation therapy.
* Evidence or history of malignant neoplasm (clinical, laboratory or imaging) except for successfully excised basal cell or squamous cell carcinoma, or successfully excised early melanoma of the skin. Subjects, who had successful tumor resection or radio-chemotherapy of breast cancer more than 10 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study. Subjects, who had successful tumor resection or radio-chemotherapy of all other tumor types and have been in remission for more than 5 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study. A dermatological exam will have ruled out any skin cancer.
* Subjects who have proliferative retinopathy, or moderate or severe non-proliferative retinopathy, from any cause (ETDRS Score > 35), clinically significant macular oedema or previous panretinal photocoagulation therapy.
* Subjects with severe renal disease defined as significant renal dysfunction evidenced by an estimated creatinine clearance of <30 mL/minute (calculated using the Cockcroft Gault formula), or receiving chronic hemodialysis therapy.
* A Stroke, TIA or MI within 3 months of entry into the study.
* Subjects with known liver disease (e.g., hepatitis B or C or cirrhosis of the liver).
* A subject with HIV, AIDS, or severe uncontrolled ulcerative colitis or Crohn's disease.
* Subjects with a current, uncorrected history of alcohol or substance abuse.
* Subjects that have been administered rhPDGF (e.g, becaplermin) or other growth factors locally within one month of randomization.
* Subjects who have received another investigational drug within 30 days of randomization or have previously received any gene transfer therapy within 3 years of entering the study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Powell, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were enrolled at a single clinical site.
Period: Overall Study
Arm/Group | AMG0001
Started | 10
Completed Month 18 Clinic Visit | 5
Completed Month 36 LTFU Questionnaire | 3
Completed | 3
Not Completed | 7
Not completed — Major amputation of index limb | 2
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | AMG0001
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Weight (kg) [Mean (Standard Deviation); unit: kg] | 81.58 (11.052)
Height (cm) [Mean (Standard Deviation); unit: cm] | 171.70 (5.921)
Past Tobacco Use [Count of Participants; unit: Participants]
  Yes - Smoking | 10
  No | 0
Current Tobacco Use [Count of Participants; unit: Participants]
  Yes - Smoking | 1
  No | 9
Alcohol Use [Count of Participants; unit: Participants]
  Yes - 1 to 2 drinks per day or less | 5
  Yes - 3 drinks per day or more | 1
  No | 4
Mobility [Count of Participants; unit: Participants]
  None | 0
  Some | 7
  Confined | 1
  Missing | 2
Ability to Self-care [Count of Participants; unit: Participants]
  None | 5
  Some | 4
  Unable | 0
  Missing | 1
Anxiety/Depression [Count of Participants; unit: Participants]
  None | 4
  Moderate | 5
  Extreme | 0
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Suspected to be Related to Injections of AMG0001
Description: All summaries and analyses will be presented in tabular or graphical form. The study is not powered for the statistical inference and the test will be considered to be descriptive.
  Treatment-emergent adverse events (TEAEs) was evaluated, and a table showing the number and percentage of subjects with occurrences categorized by System Organ Class and Preferred Term was provided by causality (relationship to study drug).
Time Frame: 18 months
Population: Not every subject analyzed may experience an adverse event likely related or possibly related to injections of AMG0001; therefore, the subject counts in the categories do not always add up to the total number analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 10
Participants
  General disorders & admin site conditions (Mild) | 1
  Infections and infestations (Mild) | 1
  Investigations (Moderate) | 1
  Eye disorders (Moderate) | 1
  Vascular disorders (Severe) | 1
  Neoplasms benign, malignant, unspecified (Severe) | 1

2. Primary Outcome: Number of Participants Discontinued Due to AEs From the Injections of AMG0001
Description: All summaries and analyses will be presented in tabular or graphical form. The study is not powered for the statistical inference and the test will be considered to be descriptive.
  Treatment-emergent adverse events (TEAEs) was evaluated, and a table showing the number and percentage of subjects with occurrences categorized by System Organ Class and Preferred Term was provided by whether the AE led to discontinuation.
Time Frame: up to 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 10
Participants
  Macular edema (likely unrelated) | 1
  Uterine leiomyosarcoma (possibly related) | 1

3. Secondary Outcome: Number of Participants in Whom the Largest Ulcer Healed Completely or Gets Smaller (Photo Confirmation)
Description: All summaries and analyses will be presented in tabular or graphical form. The study is not powered for the statistical inference and the test will be considered to be descriptive.
  A table showing the number of subjects completely healed in the target ulcer was provided at up to 6 months, > 6 months to 12 months, from >12 months to 18 months.
Time Frame: 18 Months
Population: 4 subjects classified as Rutherford Class 5 at Baseline had available data through Month 6; 1 subject through Month 12; 0 subject through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 4
Participants
  Day 0 to Month 6 | 0
  Month 6 to Month 12: number analyzed (Participants) | 1
  Month 6 to Month 12 | 0
  Month 12 to Month 18: number analyzed (Participants) | 0
  Month 12 to Month 18 | 0

4. Secondary Outcome: Number of Participants in Whom Rest Pain (Based on 10 cm VAS Scale) Reduces by 20 mm (2 cm) or More or Was Completely Relieved.
Description: All summaries and analyses will be presented in tabular or graphical form. The study is not powered for the statistical inference and the test will be considered to be descriptive.
  The severity of rest pain (based on the average over previous 7 days) recorded using the 10 cm visual analog scale (VAS).
  VAS is a 10-cm line (with score ranges 0 to 10), oriented horizontally; the left end of the line (0 mark) indicates "no pain"; the right end indicates "pain as bad as it can be."
  1. The subject is asked to mark a place on the line corresponding to the average pain intensity experienced in the last 7 days.
  2. The distance along the scale is converted into a numeric reading by measuring the distance of the subjects mark in cm from the beginning of the scale (the 0 mark).
Time Frame: 18 months
Population: 8 subjects had available data through Month 6; 6 subjects through Month 12; 4 subjects through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 8
Participants
  Day 0 to Month 6 | 1
  Month 6 to Month 12: number analyzed (Participants) | 6
  Month 6 to Month 12 | 2
  Month 12 to Month 18: number analyzed (Participants) | 4
  Month 12 to Month 18 | 2

5. Secondary Outcome: Change From Baseline of VascuQol Score for the Index Limb by Visit
Description: The VascuQol contains 5 domains (pain, symptom, activities, social, and emotional functioning); responses were scored from 0 (lowest QOL, death) to 7 (best QOL, maximum health).
  Responses were averaged for composite overall and domain-specific scores, giving equal weight to each question and domain. The composite overall is the average of domain-specific scores.
  Responses after revascularization or major amputation were included in the analysis. In the event of death, subjects were scored as 0. For the effect of treatment on individual domains, pain, symptoms, and activities were considered the most important of the 5 domains.
Time Frame: 18 months
Population: At each visit, only subjects who had a non-missing value at both baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMG0001
Number analyzed (Participants) | 8
score on a scale
  Overall (LOCF) | 0.58 (1.567)
  Activity (LOCF) | 0.54 (1.562)
  Emotional (LOCF) | 0.52 (0.935)
  Pain (LOCF) | 0.71 (2.610)
  Social (LOCF) | 0.75 (1.488)
  Symptom (LOCF) | 0.58 (2.055)
Statistical Analysis 1: Comparison: AMG0001; Overall (LOCF); Test type: Superiority; p = 0.331, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Activity (LOCF); Test type: Superiority; p = 0.362, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Emotional (LOCF); Test type: Superiority; p = 0.159, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Pain (LOCF); Test type: Superiority; p = 0.468, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Social (LOCF); Test type: Superiority; p = 0.197, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Symptom (LOCF); Test type: Superiority; p = 0.448, t-test, 2 sided

6. Secondary Outcome: Change in Hemodynamic Measurements of Change From Baseline Value of Toe Systolic Pressure (mmHg)
Description: Summary statistics was provided for baseline and change from baseline for toe systolic pressure by visit. At each visit, only subjects who have a non-missing value at both baseline and the specific visit was summarized. Two-sided one-sample t-test was performed for each visit and last observation carried forward (LOCF).
Time Frame: 18 months
Population: At each visit, only subjects who have non-missing values both at baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AMG0001
Number analyzed (Participants) | 6
mmHg
  Change from Baseline at Month 3: number analyzed (Participants) | 4
  Change from Baseline at Month 3 | 0.5 (11.96)
  Change from Baseline at Month 6 | 3.7 (12.60)
  Change from Baseline at Month 9: number analyzed (Participants) | 4
  Change from Baseline at Month 9 | 5.5 (13.48)
  Change from Baseline at Month 12: number analyzed (Participants) | 5
  Change from Baseline at Month 12 | 4.2 (9.12)
  Change from Baseline at Month 15: number analyzed (Participants) | 3
  Change from Baseline at Month 15 | 6.7 (7.37)
  Change from Baseline at Month 18: number analyzed (Participants) | 4
  Change from Baseline at Month 18 | 19.8 (13.33)
  Change from Baseline at LOCF | 16.0 (12.05)
Statistical Analysis 1: Comparison: AMG0001; Change from Baseline at Month 3; Test type: Superiority; p = 0.939, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Change from Baseline at Month 6; Test type: Superiority; p = 0.508, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Change from Baseline at Month 9; Test type: Superiority; p = 0.474, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Change from Baseline at Month 12; Test type: Superiority; p = 0.361, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Change from Baseline at Month 15; Test type: Superiority; p = 0.258, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Change from baseline at Month 18; Test type: Superiority; p = 0.059, t-test, 2 sided
Statistical Analysis 7: Comparison: AMG0001; Change from Baseline at LOCF; Test type: Superiority; p = 0.023, t-test, 2 sided

7. Secondary Outcome: Change in Hemodynamic Measurements of Change From Baseline Value of Ankle Systolic Pressure (mmHg) of the Index Leg by Visit
Description: Summary statistics was provided for baseline and change from baseline for ankle systolic pressure by visit. At each visit, only subjects who have a non-missing value at both baseline and the specific visit was summarized. Two-sided one-sample t-test was performed for each visit and last observation carried forward (LOCF).
Time Frame: 18 months
Population: At each visit, only subjects who have non-missing values both at baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AMG0001
Number analyzed (Participants) | 6
mmHg
  Change from Baseline at Month 3 (Dorsalis pedis): number analyzed (Participants) | 4
  Change from Baseline at Month 3 (Dorsalis pedis) | 10.8 (43.50)
  Change from Baseline at Month 6 (Dorsalis pedis) | 40.7 (88.18)
  Change from Baseline at Month 9 (Dorsalis pedis): number analyzed (Participants) | 5
  Change from Baseline at Month 9 (Dorsalis pedis) | 27.6 (58.12)
  Change from Baseline at Month 12 (Dorsalis pedis): number analyzed (Participants) | 4
  Change from Baseline at Month 12 (Dorsalis pedis) | 11.5 (30.16)
  Change from Baseline at Month 15 (Dorsalis pedis): number analyzed (Participants) | 3
  Change from Baseline at Month 15 (Dorsalis pedis) | -13.3 (31.13)
  Change from Baseline at Month 18 (Dorsalis pedis): number analyzed (Participants) | 3
  Change from Baseline at Month 18 (Dorsalis pedis) | 31.3 (22.81)
  Change from Baseline at LOCF (Dorsalis pedis) | 55.0 (39.07)
  Change from Baseline at Month 3 (Posterior tibial): number analyzed (Participants) | 4
  Change from Baseline at Month 3 (Posterior tibial) | 10.5 (52.45)
  Change from Baseline at Month 6 (Posterior tibial): number analyzed (Participants) | 4
  Change from Baseline at Month 6 (Posterior tibial) | -4.8 (18.41)
  Change from Baseline at Month 9 (Posterior tibial): number analyzed (Participants) | 5
  Change from Baseline at Month 9 (Posterior tibial) | -8.0 (25.02)
  Change from Baseline at Month 12 (Posterior tibial: number analyzed (Participants) | 4
  Change from Baseline at Month 12 (Posterior tibial | 2.8 (20.76)
  Change from Baseline at Month 15 (Posterior tibial: number analyzed (Participants) | 3
  Change from Baseline at Month 15 (Posterior tibial | -14.3 (23.18)
  Change from Baseline at Month 18 (Posterior tibial: number analyzed (Participants) | 3
  Change from Baseline at Month 18 (Posterior tibial | 36.7 (29.28)
  Change from Baseline at LOCF (Posterior tibial): number analyzed (Participants) | 3
  Change from Baseline at LOCF (Posterior tibial) | 19.8 (33.66)
Statistical Analysis 1: Comparison: AMG0001; Change from Baseline at Month 3 (Dorsalis pedis); Test type: Superiority; p = 0.655, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Change from Baseline at Month 6 (Dorsalis pedis); Test type: Superiority; p = 0.310, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Change from Baseline at Month 9 (Dorsalis pedis); Test type: Superiority; p = 0.348, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Change from Baseline at Month 12 (Dorsalis pedis); Test type: Superiority; p = 0.501, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Change from Baseline at Month 15 (Dorsalis pedis); Test type: Superiority; p = 0.536, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Change from Baseline at Month 18 (Dorsalis pedis); Test type: Superiority; p = 0.140, t-test, 2 sided
Statistical Analysis 7: Comparison: AMG0001; Change from Baseline at LOCF (Dorsalis pedis); Test type: Superiority; p = 0.018, t-test, 2 sided
Statistical Analysis 8: Comparison: AMG0001; Change from baseline at Month 3 (Posterior tibial); Test type: Superiority; p = 0.716, t-test, 2 sided
Statistical Analysis 9: Comparison: AMG0001; Change from baseline at Month 6 (Posterior tibial); Test type: Superiority; p = 0.641, t-test, 2 sided
Statistical Analysis 10: Comparison: AMG0001; Change from baseline at Month 9 (Posterior tibial); Test type: Superiority; p = 0.514, t-test, 2 sided
Statistical Analysis 11: Comparison: AMG0001; Change from baseline at Month 12 (Posterior tibial); Test type: Superiority; p = 0.808, t-test, 2 sided
Statistical Analysis 12: Comparison: AMG0001; Change from baseline at Month 15 (Posterior tibial); Test type: Superiority; p = 0.396, t-test, 2 sided
Statistical Analysis 13: Comparison: AMG0001; Change from baseline at Month 18 (Posterior tibial); Test type: Superiority; p = 0.162, t-test, 2 sided
Statistical Analysis 14: Comparison: AMG0001; Change from baseline at LOCF (Posterior tibial); Test type: Superiority; p = 0.259, t-test, 2 sided

8. Secondary Outcome: Change in Hemodynamic Measurements of Change From Baseline Value of Brachial Systolic Pressure (mmHg)
Description: Summary statistics was provided for baseline and change from baseline for right/left brachial systolic pressure by visit. At each visit, only subjects who have a non-missing value at both baseline and the specific visit was summarized. Two-sided one-sample t-test was performed for each visit and last observation carried forward (LOCF).
Time Frame: 18 months
Population: At each visit, only subjects who have non-missing values both at baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AMG0001
Number analyzed (Participants) | 8
mmHg
  Change from Baseline at Month 3 (Right): number analyzed (Participants) | 6
  Change from Baseline at Month 3 (Right) | -4.5 (24.42)
  Change from Baseline at Month 6 (Right): number analyzed (Participants) | 7
  Change from Baseline at Month 6 (Right) | -1.1 (30.80)
  Change from Baseline at Month 9 (Right): number analyzed (Participants) | 5
  Change from Baseline at Month 9 (Right) | -4.2 (13.12)
  Change from Baseline at Month 12 (Right): number analyzed (Participants) | 5
  Change from Baseline at Month 12 (Right) | -9.6 (18.12)
  Change from Baseline at Month 15 (Right): number analyzed (Participants) | 4
  Change from Baseline at Month 15 (Right) | -4.3 (8.14)
  Change from Baseline at Month 18 (Right): number analyzed (Participants) | 4
  Change from Baseline at Month 18 (Right) | 5.8 (15.22)
  Change from Baseline at LOCF (Right) | 12.5 (20.91)
  Change from Baseline at Month 3 (Left): number analyzed (Participants) | 7
  Change from Baseline at Month 3 (Left) | -10.9 (18.67)
  Change from Baseline at Month 6 (Left): number analyzed (Participants) | 6
  Change from Baseline at Month 6 (Left) | -7.8 (20.52)
  Change from Baseline at Month 9 (Left): number analyzed (Participants) | 5
  Change from Baseline at Month 9 (Left) | -0.6 (13.90)
  Change from Baseline at Month 12 (Left): number analyzed (Participants) | 5
  Change from Baseline at Month 12 (Left) | -6.6 (16.79)
  Change from Baseline at Month 15 (Left): number analyzed (Participants) | 4
  Change from Baseline at Month 15 (Left) | 1.0 (15.77)
  Change from Baseline at Month 18 (Left): number analyzed (Participants) | 4
  Change from Baseline at Month 18 (Left) | 8.3 (13.20)
  Change from Baseline at LOCF (Left) | 6.6 (13.70)
Statistical Analysis 1: Comparison: AMG0001; Change from Baseline at Month 3; Test type: Superiority; p = 0.671, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Change from Baseline at Month 6; Test type: Superiority; p = 0.925, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Change from Baseline at Month 9; Test type: Superiority; p = 0.514, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Change from Baseline at Month 12; Test type: Superiority; p = 0.302, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Change from Baseline at Month 15; Test type: Superiority; p = 0.373, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Change from Baseline at Month 18; Test type: Superiority; p = 0.505, t-test, 2 sided
Statistical Analysis 7: Comparison: AMG0001; Change from Baseline at LOCF; Test type: Superiority; p = 0.135, t-test, 2 sided
Statistical Analysis 8: Comparison: AMG0001; Change from baseline at month 3 (Left); Test type: Superiority; p = 0.175, t-test, 2 sided
Statistical Analysis 9: Comparison: AMG0001; Change from baseline at month 6 (Left); Test type: Superiority; p = 0.393, t-test, 2 sided
Statistical Analysis 10: Comparison: AMG0001; Change from baseline at month 9 (Left); Test type: Superiority; p = 0.928, t-test, 2 sided
Statistical Analysis 11: Comparison: AMG0001; Change from baseline at month 12 (Left); Test type: Superiority; p = 0.429, t-test, 2 sided
Statistical Analysis 12: Comparison: AMG0001; Change from baseline at month 15 (Left); Test type: Superiority; p = 0.907, t-test, 2 sided
Statistical Analysis 13: Comparison: AMG0001; Change from baseline at month 18 (Left); Test type: Superiority; p = 0.300, t-test, 2 sided
Statistical Analysis 14: Comparison: AMG0001; Change from baseline at LOCF (Left); Test type: Superiority; p = 0.214, t-test, 2 sided

9. Secondary Outcome: Change in Hemodynamic Measurement of Baseline Calculated Toe Brachial Index (TBI) of the Index Leg by Visit
Description: Summary statistics was provided for baseline and change from baseline for toe brachial index (TBI) by visit. At each visit, only subjects who have a non-missing value at both baseline and the specific visit was summarized. Two-sided one-sample t-test was performed for each visit and last observation carried forward (LOCF).
  TBI was calculated by dividing the toe systolic blood pressure by the brachial systolic blood pressure. TBI was calculated at baseline and at each visit. The change in TBI at each visit compared to the baseline value was recorded.
Time Frame: 18 months
Population: At each visit, only subjects who have non-missing values both at baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AMG0001
Number analyzed (Participants) | 6
ratio
  Change from Baseline at Month 3: number analyzed (Participants) | 4
  Change from Baseline at Month 3 | 0.0180 (0.0709)
  Change from Baseline at Month 6 | 0.040 (0.0710)
  Change from Baseline at Month 9: number analyzed (Participants) | 4
  Change from Baseline at Month 9 | 0.040 (0.0779)
  Change from Baseline at Month 12: number analyzed (Participants) | 5
  Change from Baseline at Month 12 | 0.044 (0.0619)
  Change from Baseline at Month 15: number analyzed (Participants) | 3
  Change from Baseline at Month 15 | 0.060 (0.0557)
  Change from Baseline at Month 18: number analyzed (Participants) | 4
  Change from Baseline at Month 18 | 0.123 (0.0907)
  Change from Baseline at LOCF | 0.095 (0.0831)
Statistical Analysis 1: Comparison: AMG0001; Change from Baseline at Month 3; Test type: Superiority; p = 0.655, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Change from Baseline at Month 6; Test type: Superiority; p = 0.226, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Change from Baseline at Month 9; Test type: Superiority; p = 0.380, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Change from Baseline at Month 12; Test type: Superiority; p = 0.187, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Change from Baseline at Month 15; Test type: Superiority; p = 0.203, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Change from Baseline at Month 18; Test type: Superiority; p = 0.074, t-test, 2 sided
Statistical Analysis 7: Comparison: AMG0001; Change from Baseline at LOCF; Test type: Superiority; p = 0.038, t-test, 2 sided

10. Secondary Outcome: Change in Hemodynamic Measurement of Baseline Calculated ABI of the Index Leg by Visit
Description: Summary statistics was provided for baseline and change from baseline for ankle brachial index (ABI) by visit. At each visit, only subjects who have a non-missing value at both baseline and the specific visit was summarized. Two-sided one-sample t-test was performed for each visit and last observation carried forward (LOCF).
  ABI was calculated by dividing the ankle systolic blood pressure by the brachial systolic blood pressure. ABI was calculated at baseline and at each visit. The change in ABI at each visit compared to the baseline value was recorded.
Time Frame: 18 months
Population: At each visit, only subjects who have non-missing values both at baseline and the specific visit was summarized.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AMG0001
Number analyzed (Participants) | 7
ratio
  Change from Baseline at Month 3: number analyzed (Participants) | 5
  Change from Baseline at Month 3 | 0.286 (0.4711)
  Change from Baseline at Month 6: number analyzed (Participants) | 6
  Change from Baseline at Month 6 | 0.115 (0.3642)
  Change from Baseline at Month 9: number analyzed (Participants) | 5
  Change from Baseline at Month 9 | 0.102 (0.2395)
  Change from Baseline at Month 12: number analyzed (Participants) | 5
  Change from Baseline at Month 12 | 0.254 (0.3909)
  Change from Baseline at Month 15: number analyzed (Participants) | 3
  Change from Baseline at Month 15 | -0.097 (0.1815)
  Change from Baseline at Month 18: number analyzed (Participants) | 3
  Change from Baseline at Month 18 | 0.210 (0.1709)
  Change from Baseline at LOCF | 0.431 (0.3365)
Statistical Analysis 1: Comparison: AMG0001; Change from Baseline at Month 3; Test type: Superiority; p = 0.246, t-test, 2 sided
Statistical Analysis 2: Comparison: AMG0001; Change from Baseline at Month 6; Test type: Superiority; p = 0.474, t-test, 2 sided
Statistical Analysis 3: Comparison: AMG0001; Change from Baseline at Month 9; Test type: Superiority; p = 0.395, t-test, 2 sided
Statistical Analysis 4: Comparison: AMG0001; Change from Baseline at Month 12; Test type: Superiority; p = 0.220, t-test, 2 sided
Statistical Analysis 5: Comparison: AMG0001; Change from Baseline at Month 15; Test type: Superiority; p = 0.454, t-test, 2 sided
Statistical Analysis 6: Comparison: AMG0001; Change from Baseline at Month 18; Test type: Superiority; p = 0.167, t-test, 2 sided
Statistical Analysis 7: Comparison: AMG0001; Change from Baseline at LOCF; Test type: Superiority; p = 0.015, t-test, 2 sided

11. Secondary Outcome: Subjects Who Had Myocardial Infarction (MI), Stroke, Major Amputation, Revascularization (by Surgical Bypass, Endovascular Intervention, Hybrid Procedure), or All-cause Death
Description: A summary table including counts and percentages was provided for subjects who had MI, stroke, major amputation, revascularization, or all-cause death for the time periods: 0 to Month 6, 0 to Month 12, 0 to Month 18.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 10
Participants
  Month 0 to 6: Myocardial infarction | 0
  Month 0 to 6: Stroke | 0
  Month 0 to 6: Major amputation of the index leg | 1
  Month 0 to 6: Revascularization of the index leg | 1
  Month 0 to 6: All-cause death | 1
  Month 0 to 6: No events recorded | 7
  Month 0 to 12: Myocardial infarction | 0
  Month 0 to 12: Stroke | 0
  Month 0 to 12: Major amputation of the index leg | 2
  Month 0 to 12: Revascularization of the index leg | 1
  Month 0 to 12: All-cause death | 2
  Month 0 to 12: No events recorded | 5
  Month 0 to 18: Myocardial infarction | 0
  Month 0 to 18: Stroke | 0
  Month 0 to 18: Major amputation of the index leg | 2
  Month 0 to 18: Revascularization of the index leg | 3
  Month 0 to 18: All-cause death | 3
  Month 0 to 18: No events recorded | 2

12. Secondary Outcome: Number of Participants With Worsening CLI Event of Index Leg
Description: A summary table and listing of worsening CLI-related events of the index leg including any new or worsening events, worsening rest pain, new ulcer or worsening ulcer, new or worsening wound infection, peripheral vascular intervention, complication of a peripheral vascular intervention, cellulitis, and amputation due to worsening CLI was provided.
Time Frame: 18 months
Population: Number analyzed in one or more rows differs from overall number analyzed due to subject study discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 7
Participants
  Up to 3M : Any CLI-related events | 3
  Up to 3M : Worsening rest pain | 3
  Up to 3M : New ulcer | 2
  Up to 3M : Wound infection (new or worsening) | 1
  Up to 3M : Amputation due to Worsening CLI | 1
  Up to 3M : Peripheral vascular intervention | 1
  Up to 3M : Complication vascular intervention | 0
  Up to 3M : Cellulitis | 1
  Up to 3M : Worsening of ulcer | 1
  3M to 6M : Any CLI-related events | 2
  3M to 6M : Worsening rest pain | 2
  3M to 6M : New ulcer | 2
  3M to 6M : Wound infection (new or worsening) | 0
  3M to 6M : Amputation due to Worsening CLI | 0
  3M to 6M : Peripheral vascular intervention | 0
  3M to 6M : Complication of vascular intervention | 0
  3M to 6M : Cellulitis | 0
  3M to 6M : Worsening of ulcer | 1
  6M to 9M : Any CLI-related events: number analyzed (Participants) | 6
  6M to 9M : Any CLI-related events | 2
  6M to 9M : Worsening rest pain: number analyzed (Participants) | 6
  6M to 9M : Worsening rest pain | 0
  6M to 9M : New ulcer: number analyzed (Participants) | 6
  6M to 9M : New ulcer | 0
  6M to 9M : Wound infection (new or worsening): number analyzed (Participants) | 6
  6M to 9M : Wound infection (new or worsening) | 1
  Month 6 up to 9 : Amputation due to Worsening CLI: number analyzed (Participants) | 6
  Month 6 up to 9 : Amputation due to Worsening CLI | 2
  Month 6 up to 9 : Peripheral vascular intervention: number analyzed (Participants) | 6
  Month 6 up to 9 : Peripheral vascular intervention | 0
  6M to 9M : Complication of vascular intervention: number analyzed (Participants) | 6
  6M to 9M : Complication of vascular intervention | 0
  Month 6 up to 9 : Cellulitis: number analyzed (Participants) | 6
  Month 6 up to 9 : Cellulitis | 0
  Month 6 up to 9 : Worsening of ulcer: number analyzed (Participants) | 6
  Month 6 up to 9 : Worsening of ulcer | 0
  9M to 12M : Any CLI-related events: number analyzed (Participants) | 6
  9M to 12M : Any CLI-related events | 1
  Month 9 up to 12 : Worsening rest pain: number analyzed (Participants) | 6
  Month 9 up to 12 : Worsening rest pain | 0
  Month 9 up to 12 : New ulcer: number analyzed (Participants) | 6
  Month 9 up to 12 : New ulcer | 0
  9M to 12M : Wound infection (new or worsening): number analyzed (Participants) | 6
  9M to 12M : Wound infection (new or worsening) | 0
  Month 9 up to 12 : Amputation due to Worsening CLI: number analyzed (Participants) | 6
  Month 9 up to 12 : Amputation due to Worsening CLI | 1
  9M to 12M : Peripheral vascular intervention: number analyzed (Participants) | 6
  9M to 12M : Peripheral vascular intervention | 0
  9M to 12M : Complication of vascular intervention: number analyzed (Participants) | 6
  9M to 12M : Complication of vascular intervention | 0
  Month 9 up to 12 : Cellulitis: number analyzed (Participants) | 6
  Month 9 up to 12 : Cellulitis | 0
  Month 9 up to 12 : Worsening of ulcer: number analyzed (Participants) | 6
  Month 9 up to 12 : Worsening of ulcer | 0
  12M to 15M : Any CLI-related events: number analyzed (Participants) | 5
  12M to 15M : Any CLI-related events | 2
  Month 12 up to 15 : Worsening rest pain: number analyzed (Participants) | 5
  Month 12 up to 15 : Worsening rest pain | 0
  Month 12 up to 15 : New ulcer: number analyzed (Participants) | 5
  Month 12 up to 15 : New ulcer | 0
  12M to 15M : Wound infection (new or worsening): number analyzed (Participants) | 5
  12M to 15M : Wound infection (new or worsening) | 1
  12M to 15M : Amputation due to Worsening CLI: number analyzed (Participants) | 5
  12M to 15M : Amputation due to Worsening CLI | 0
  12M to 15M : Peripheral vascular intervention: number analyzed (Participants) | 5
  12M to 15M : Peripheral vascular intervention | 1
  12M to 15M : Complication of vascular intervention: number analyzed (Participants) | 5
  12M to 15M : Complication of vascular intervention | 0
  Month 12 up to 15 : Cellulitis: number analyzed (Participants) | 5
  Month 12 up to 15 : Cellulitis | 0
  Month 12 up to 15 : Worsening of ulcer: number analyzed (Participants) | 5
  Month 12 up to 15 : Worsening of ulcer | 0
  15M to 18M : Any CLI-related events: number analyzed (Participants) | 5
  15M to 18M : Any CLI-related events | 2
  Month 15 up to 18 : Worsening rest pain: number analyzed (Participants) | 5
  Month 15 up to 18 : Worsening rest pain | 1
  Month 15 up to 18 : New ulcer: number analyzed (Participants) | 5
  Month 15 up to 18 : New ulcer | 0
  15M to 18M : Wound infection (new or worsening): number analyzed (Participants) | 5
  15M to 18M : Wound infection (new or worsening) | 0
  15M to 18M : Amputation due to Worsening CLI: number analyzed (Participants) | 5
  15M to 18M : Amputation due to Worsening CLI | 1
  15M to 18M : Peripheral vascular intervention: number analyzed (Participants) | 5
  15M to 18M : Peripheral vascular intervention | 1
  15M to 18M : Complication of vascular intervention: number analyzed (Participants) | 5
  15M to 18M : Complication of vascular intervention | 0
  Month 15 up to 18 : Cellulitis: number analyzed (Participants) | 5
  Month 15 up to 18 : Cellulitis | 0
  Month 15 up to 18 : Worsening of ulcer: number analyzed (Participants) | 5
  Month 15 up to 18 : Worsening of ulcer | 0

13. Secondary Outcome: Number of Participants With Shift From Baseline in Rutherford Classification
Description: Shift from baseline in Rutherford classification was summarized by study visit. Patients enrolled in the study were classified as either Rutherford 4 or Rutherford 5 at baseline.
  Rutherford category (clinical description) 0 (Asymptomatic - no hemodynamically significant occlusive disease)
  1. (Mild claudication)
  2. (Moderate claudication)
  3. (Severe claudication)
  4. (Ischemic rest pain)
  5. (Minor tissue loss - nonhealing ulcer, focal gangrene with diffuse pedal ischemia)
  6. (Major tissue loss - extending above TM level, functional foot no longer salvageable)
Time Frame: 18 months
Population: Number analyzed in one or more rows differs from overall number analyzed due to subject study discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG0001
Number analyzed (Participants) | 5
Participants
  Up to Month 3 (Baseline R4): Shift to R1 | 0
  Up to Month 3 (Baseline R4): Shift to R2 | 0
  Up to Month 3 (Baseline R4): Shift to R3 | 0
  Up to Month 3 (Baseline R4): Shift to R4 | 4
  Up to Month 3 (Baseline R4): Shift to R5 | 1
  Up to Month 3 (Baseline R4): Shift to R6 | 0
  Up to Month 3 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 0
  Month 3 to 6 (Baseline R4): number analyzed (Participants) | 4
  Month 3 to 6 (Baseline R4): Shift to R1 | 0
  Month 3 to 6 (Baseline R4): Shift to R2 | 0
  Month 3 to 6 (Baseline R4): Shift to R3 | 1
  Month 3 to 6 (Baseline R4): Shift to R4 | 2
  Month 3 to 6 (Baseline R4): Shift to R5 | 1
  Month 3 to 6 (Baseline R4): Shift to R6 | 0
  Month 3 to 6 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 0
  Month 6 to 9 (Baseline R4): number analyzed (Participants) | 2
  Month 6 to 9 (Baseline R4): Shift to R1 | 0
  Month 6 to 9 (Baseline R4): Shift to R2 | 1
  Month 6 to 9 (Baseline R4): Shift to R3 | 1
  Month 6 to 9 (Baseline R4): Shift to R4 | 0
  Month 6 to 9 (Baseline R4): Shift to R5 | 0
  Month 6 to 9 (Baseline R4): Shift to R6 | 0
  Month 6 to 9 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 0
  Month 9 to 12 (Baseline R4): number analyzed (Participants) | 4
  Month 9 to 12 (Baseline R4): Shift to R1 | 1
  Month 9 to 12 (Baseline R4): Shift to R2 | 0
  Month 9 to 12 (Baseline R4): Shift to R3 | 1
  Month 9 to 12 (Baseline R4): Shift to R4 | 1
  Month 9 to 12 (Baseline R4): Shift to R5 | 1
  Month 9 to 12 (Baseline R4): Shift to R6 | 0
  Month 9 to 12 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 0
  Month 12 to 15 (Baseline R4): number analyzed (Participants) | 4
  Month 12 to 15 (Baseline R4): Shift to R1 | 0
  Month 12 to 15 (Baseline R4): Shift to R2 | 1
  Month 12 to 15 (Baseline R4): Shift to R3 | 0
  Month 12 to 15 (Baseline R4): Shift to R4 | 1
  Month 12 to 15 (Baseline R4): Shift to R5 | 1
  Month 12 to 15 (Baseline R4): Shift to R6 | 0
  Month 12 to 15 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 1
  Month 15 to 18 (Baseline R4): number analyzed (Participants) | 4
  Month 15 to 18 (Baseline R4): Shift to R1 | 0
  Month 15 to 18 (Baseline R4): Shift to R2 | 0
  Month 15 to 18 (Baseline R4): Shift to R3 | 2
  Month 15 to 18 (Baseline R4): Shift to R4 | 1
  Month 15 to 18 (Baseline R4): Shift to R5 | 1
  Month 15 to 18 (Baseline R4): Shift to R6 | 0
  Month 15 to 18 (Baseline R4): Discontinuation due to Death, AE or CLI Event | 0
  Up to Month 3 (Baseline R5): number analyzed (Participants) | 4
  Up to Month 3 (Baseline R5): Shift to R1 | 0
  Up to Month 3 (Baseline R5): Shift to R2 | 0
  Up to Month 3 (Baseline R5): Shift to R3 | 0
  Up to Month 3 (Baseline R5): Shift to R4 | 0
  Up to Month 3 (Baseline R5): Shift to R5 | 3
  Up to Month 3 (Baseline R5): Shift to R6 | 0
  Up to Month 3 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 1
  Month 3 to 6 (Baseline R5): number analyzed (Participants) | 3
  Month 3 to 6 (Baseline R5): Shift to R1 | 0
  Month 3 to 6 (Baseline R5): Shift to R2 | 0
  Month 3 to 6 (Baseline R5): Shift to R3 | 0
  Month 3 to 6 (Baseline R5): Shift to R4 | 0
  Month 3 to 6 (Baseline R5): Shift to R5 | 2
  Month 3 to 6 (Baseline R5): Shift to R6 | 0
  Month 3 to 6 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 1
  Month 6 to 9 (Baseline R5): number analyzed (Participants) | 2
  Month 6 to 9 (Baseline R5): Shift to R1 | 0
  Month 6 to 9 (Baseline R5): Shift to R2 | 0
  Month 6 to 9 (Baseline R5): Shift to R3 | 0
  Month 6 to 9 (Baseline R5): Shift to R4 | 0
  Month 6 to 9 (Baseline R5): Shift to R5 | 2
  Month 6 to 9 (Baseline R5): Shift to R6 | 0
  Month 6 to 9 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 0
  Month 9 to 12 (Baseline R5): number analyzed (Participants) | 2
  Month 9 to 12 (Baseline R5): Shift to R1 | 0
  Month 9 to 12 (Baseline R5): Shift to R2 | 0
  Month 9 to 12 (Baseline R5): Shift to R3 | 0
  Month 9 to 12 (Baseline R5): Shift to R4 | 0
  Month 9 to 12 (Baseline R5): Shift to R5 | 0
  Month 9 to 12 (Baseline R5): Shift to R6 | 0
  Month 9 to 12 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 2
  Month 12 to 15 (Baseline R5): number analyzed (Participants) | 0
  Month 12 to 15 (Baseline R5): Shift to R1 | 0
  Month 12 to 15 (Baseline R5): Shift to R2 | 0
  Month 12 to 15 (Baseline R5): Shift to R3 | 0
  Month 12 to 15 (Baseline R5): Shift to R4 | 0
  Month 12 to 15 (Baseline R5): Shift to R5 | 0
  Month 12 to 15 (Baseline R5): Shift to R6 | 0
  Month 12 to 15 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 0
  Month 15 to 18 (Baseline R5): number analyzed (Participants) | 0
  Month 15 to 18 (Baseline R5): Shift to R1 | 0
  Month 15 to 18 (Baseline R5): Shift to R2 | 0
  Month 15 to 18 (Baseline R5): Shift to R3 | 0
  Month 15 to 18 (Baseline R5): Shift to R4 | 0
  Month 15 to 18 (Baseline R5): Shift to R5 | 0
  Month 15 to 18 (Baseline R5): Shift to R6 | 0
  Month 15 to 18 (Baseline R5): Discontinuation due to Death, AE or CLI Event | 0

ADVERSE EVENTS:
Time Frame: Adverse events were documented and followed from the start of the first dose of study product (Day 0), until the final outcome is known or until the end of the study safety follow-up period (Month 36).
Arm/Group | AMG0001
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG0001 (N=10)
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Intestinal ischemia (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Post procedural hematoma (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Leg amputation (Surgical and medical procedures) | 1
Toe amputation (Surgical and medical procedures) | 1
Ischemic limb pain (Vascular disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Uterine Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG0001 (N=10)
Administration site reaction (General disorders) | 9
Injection site discharge (General disorders) | 1
Oversensing (General disorders) | 1
Excoriation (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 2
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Anemia postoperative (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Blood blister (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Blood glucose increased (Investigations) | 2
Oxygen saturation decreased (Investigations) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myoclonus (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
anaemia (Blood and lymphatic system disorders) | 2
Diabetic retinopathy (Eye disorders) | 1
Macular oedema (Eye disorders) | 1
Vitreous adhesions (Eye disorders) | 1
hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT02016755/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02016755/SAP_001.pdf